CLINICAL TRIAL: NCT02462369
Title: The Effects of Saxagliptin 5mg, Once Daily for 52 Weeks on 24 Hour Urine Albumin Creatinine Rate(ACR) , in Patients With Type 2 Diabetes Mellitus Who Have Inadequate Glycaemic Control on Metformin or/and Acarbose
Brief Title: Saxagliptin's Effects on Microalbuminuria Improvement in Type 2 Diabetic Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: The Second Hospital of Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SecondNanjingMU
Record Dates: First submitted 2015-04-08; First posted 2015-06-04 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-04

CONDITIONS: Microalbuminuria; Microalbuminuria /Creatinine Ratios ACR
MeSH Terms: interventions — saxagliptin; glimepiride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Saxagliptin (Experimental): Saxagliptin 5mg/d, 52 weeks
  Interventions: Drug: Saxagliptin
- glimepiride (Active Comparator): glimepiride 1~4mg/d,52 weeks
  Interventions: Drug: glimepiride

INTERVENTIONS:
Drug: Saxagliptin
  Arms: Saxagliptin
Drug: glimepiride
  Arms: glimepiride

SUMMARY:
This study compare the effects on microalbuminuria improvement in type 2 diabetes mellitus (T2DM) treated with saxagliptin or glimepiride.All patients received metformin and/or acarbose, and randomly receive saxagliptin (5mg/d) or glimepiride (1-4mg/d).

DETAILED DESCRIPTION:
Both sitagliptin and glimepiride are hypoglycemic agents,but they do so by different mechanisms.sitagliptin can delay degradation of glucagon-like peptide -1 (GLP-1) by inhibit DPPIV to decrease serum glucose level.glimepiride stimulates islets B cell to secrete insulin to decrease serum glucose level.

Preclinical studies and several clinical trials (including vildagliptin, sitagliptin, linagliptin, exenatide) suggested that DPP-4i/GLP-1 might have a potential to lower albuminuria, albumin-creatinine ratio (ACR) or improve glomerular filtration rate(GFR) and the effect might be independent of changes in glucose control. Recently, SAVOR outcomes also showed that saxagliptin might have nephroprotective effects, and the proportion of patients with microalbuminuria converted into normal albuminuria after saxagliptin treatment for 1 year is 31.3%, but the mechanism is still unclear.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures
2. Diagnosed with type 2 diabetes with stable, doses of metformin (1000mg~2550mg/d) or acarbose (100mg~300mg/d) at least 60 days
3. Men and women (non-pregnant and using a medically approved birth-control method) aged at age ≥20 and ≤70 years at screening
4. HbA1c ≥ 7.0% and ≤ 9.0% at screening
5. 24-hour urinary albumin level of 30-300 mg/24 h

Exclusion Criteria:

1．Women, who are pregnant, or intending to become pregnant during the study period, currently lactating females, or women of child-bearing potential not using highly effective, medically approved birth control methods.

2. Diagnosis or history of:

* Type 1 diabetes mellitus, diabetes resulting from pancreatic injury or secondary forms of diabetes, e.g acromegaly or Cushing's syndrome.
* Acute metabolic diabetic complications such as ketoacidosis or hyperosmolar coma within the past 6 months.

  3. Previous treatment with any dipeptidyl peptidase-4 (DPP4) inhibitor or GLP-1 receptor agonists within the past 6 months． 4. History of hypersensitivity reaction (e.g., anaphylaxis, angioedema, exfoliative skin conditions) to dipeptidyl peptidase-4 inhibitor (DPP4), glimepiride, metformin or acarbose.

  5. Treatment with systemic glucocorticoids (oral, intravenous) for more than consecutive 7 days within the past 6 months.

  6. Triglycerides (fasting) > 4.5 mmol/L (> 400 mg/dL) at screening or within 4 weeks prior to screening.

  7. Patients with clinically apparent liver disease characterized by either one of the following:
* alanine aminotransferase((ALT) or aspartate aminotransferase(AST) > 3x upper limit of normal (ULN) confirmed on two consecutive measurements within 4 weeks prior to screening period
* Impaired excretory (eg, hyperbilirubinemia) and/or synthetic function, or other conditions of decompensated liver disease such as coagulopathy, hepatic encephalopathy, hypoalbuminemia, ascites and bleeding from oesophageal varices.
* Acute viral or active autoimmune, alcoholic, or other types of hepatitis.

  8. Patients with moderate /severe renal impairment or end-stage renal disease (CrCl ≤ 50 mL/min) at screening or within 4 weeks prior to screening

  9. Congestive heart failure defined as New York Heart Association (NYHA) class III or IV.

  10. Significant cardiovascular history within the past 3 months prior to screening defined as: myocardial infarction, coronary angioplasty or bypass graft(s), valvular disease or repair, unstable angina pectoris, transient ischemic attack, or cerebrovascular accident.

  11. History of chronic pancreatitis or idiopathic acute pancreatitis.

  12. History of gastrointestinal disease including gastroenterostomy, enterectomy, severe hernia, intestinal obstruction, intestinal ulcer.

  13. History of medullary thyroid carcinoma.

  14. History of alcohol abuse or illegal drug abuse within the past 12 months.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2015-06; Primary Completion 2017-04 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
microalbuminuria improvement in T2DM treated with saxagliptin | 52 weeks

SECONDARY OUTCOMES:
incidence of hypoglycaemia of saxagliptin or glimepiride | 52 weeks

REFERENCES:
- [Background] Mosenzon O, Bhatt DL, Likwat L, et al. Effect of saxagliptin on renal outcomes. 2014 ADA poster. 544-P.
- [Result] Parving HH, Lewis JB, Ravid M, Remuzzi G, Hunsicker LG; DEMAND investigators. Prevalence and risk factors for microalbuminuria in a referred cohort of type II diabetic patients: a global perspective. Kidney Int. 2006 Jun;69(11):2057-63. doi: 10.1038/sj.ki.5000377. PMID 16612330
- [Result] Phung OJ, Scholle JM, Talwar M, Coleman CI. Effect of noninsulin antidiabetic drugs added to metformin therapy on glycemic control, weight gain, and hypoglycemia in type 2 diabetes. JAMA. 2010 Apr 14;303(14):1410-8. doi: 10.1001/jama.2010.405. PMID 20388897
- [Result] Hattori S. Sitagliptin reduces albuminuria in patients with type 2 diabetes. Endocr J. 2011;58(1):69-73. doi: 10.1507/endocrj.k10e-382. Epub 2010 Dec 28. PMID 21206136
- [Result] Liu WJ, Xie SH, Liu YN, Kim W, Jin HY, Park SK, Shao YM, Park TS. Dipeptidyl peptidase IV inhibitor attenuates kidney injury in streptozotocin-induced diabetic rats. J Pharmacol Exp Ther. 2012 Feb;340(2):248-55. doi: 10.1124/jpet.111.186866. Epub 2011 Oct 24. PMID 22025647
- [Result] Groop PH, Cooper ME, Perkovic V, Emser A, Woerle HJ, von Eynatten M. Linagliptin lowers albuminuria on top of recommended standard treatment in patients with type 2 diabetes and renal dysfunction. Diabetes Care. 2013 Nov;36(11):3460-8. doi: 10.2337/dc13-0323. Epub 2013 Sep 11. PMID 24026560